CLINICAL TRIAL: NCT05263739
Title: A First-in-Human Phase I, Open Label, Multiple Dose, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of Anti-BAFFR mAb, ESG206 in Subjects With B-cell Lymphoid Malignancies
Brief Title: A First-in-Human Phase I Study of ESG206 in Subjects With B-cell Lymphoid Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Collaborators: Escugen (Australia) Biotechnology Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ESG206-101
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: B-cell Lymphoid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ESG206 dose level 1 (Experimental): ESG206 will be administered intravenously at dose level 1 every two weeks in a 28-day cycle.
  Interventions: Drug: ESG206
- ESG206 dose level 2 (Experimental): ESG206 will be administered intravenously at dose level 2 every two weeks in a 28-day cycle.
  Interventions: Drug: ESG206
- ESG206 dose level 3 (Experimental): ESG206 will be administered intravenously at dose level 3 every two weeks in a 28-day cycle.
  Interventions: Drug: ESG206
- ESG206 dose level 4 (Experimental): ESG206 will be administered intravenously at dose level 4 every two weeks in a 28-day cycle.
  Interventions: Drug: ESG206
- ESG206 dose level 5 (Experimental): ESG206 will be administered intravenously at dose level 5 every two weeks in a 28-day cycle.
  Interventions: Drug: ESG206

INTERVENTIONS:
Drug: ESG206 — Administered via intravenous (IV) infusion

SUMMARY:
This is a first-in-human phase I, multicenter, open label, sequential-cohort, dose escalation study of ESG206. The purpose is to evaluate the clinical safety, tolerability, PK, and preliminary efficacy and to establish the MTD, if any, and RP2D(s) of ESG206 in adult subjects with B lymphoid malignancies.

DETAILED DESCRIPTION:
This is a first-in-human phase I, multicenter, open label, sequential-cohort, dose escalation study of ESG206. The study will follow a modified 3+3 dose escalation scheme. Dose escalation will continue until identification of MTD or the predicted efficacy dose in the event that a MTD is not identified due to paucity of DLTs. Toxicity including dose-limiting toxicity (DLT) observed in Cycle 1 of the first 28 days will be used to determine escalation to the next dose level as described below.

Five dose levels are planned. Dose choosing will be determined by the SMC and the sponsor based on the pharmacokinetics, tolerability and preliminary antitumor activities, as well as other available data.

Subjects will be monitored for safety, tolerability, and efficacy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial.
* Male or female and at least 18 years of age.
* Subjects must have a histologically confirmed (or documented), incurable B-cell hematologic malignancy that had progressed despite standard of care therapy and for which there was no alternative therapy of proven benefit or no effective standard therapy is available or tolerable.
* Measurable or evaluable Disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject must have adequate organ function.

Exclusion Criteria:

* Has had prior chemotherapy, targeted therapy, immunotherapy or any other agents used as systemic treatment for cancer, within 14 days before first dosing.
* Had major surgery within 4 weeks before first dosing.
* Had undergone an autologous stem cell transplant within 100 days before first dosing.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, or renal disease).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product or excipients.
* Pregnant or breastfeeding women.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events | First dose date up to last dose plus 30 days
  Treatment-emergent adverse events (TEAEs) were defined as: Any AE that happens after treatment initiation,.or AE that was present at time of treatment initiation but worsened after treatment initiation, or AE that was present and resolved prior to treatment and reappeared after treatment initiation after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0.

SECONDARY OUTCOMES:
Cmax | Up to 20 months
  Maximum observed plasma concentration
AUC0-inf | Up to 20 months
  Area under the serum concentration time curve from time 0 extrapolated to infinity
Tmax | Up to 20 months
  Time to maximum plasma concentration
T1/2 | Up to 20 months
  Half-life
Overall Response (OR) | Up to 20 months
  Defined as complete response (CR) + partial response (PR)
Progression-free Survival (PFS) | Up to 20 months
  Defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression or death from any cause
ADA | Up to 20 months
  Incidence of anti-drug antibodies

IPD SHARING:
Plan to Share IPD: No